CLINICAL TRIAL: NCT01168427
Title: Reveal® In-Office Implants Study
Brief Title: Reveal In-Office Implants
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: Reveal In-Office Implants
Record Dates: First submitted 2010-07-21; First posted 2010-07-23 (Estimated); Results first posted 2012-07-26 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-01

CONDITIONS: Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Reveal® DX or Reveal® XT Insertable Cardiac Monitor — Reveal® DX and Reveal® XT Insertable Cardiac Monitors are implantable patient-activated and automatically-activated monitoring systems that record subcutaneous ECG.

SUMMARY:
The purpose of this study is to gather evidence about the safety and feasibility of performing the implant procedure for the Reveal Insertable Cardiac Monitor (ICM) in an office or clinic setting rather than the traditional hospital operating room, cardiac catheterization or electrophysiology (EP) laboratory setting.

ELIGIBILITY:
Inclusion Criteria:

* Patient is indicated for continuous arrhythmia monitoring with an Insertable Cardiac Monitor (ICM)
* Patient is willing to undergo implant in clinic setting with only local anesthetic and/or oral anti-anxiety medications for sedation
* Patient is 18 years of age or older
* Patient is willing and able to provide consent and authorize the use and disclosure of health information
* Patient is willing and able to comply with the protocol including the required follow-up

Exclusion Criteria:

* Patient has reduced immune function or is otherwise at high risk for infection
* Patient has had a recent (within 30 days) or otherwise unresolved infection
* Patient is implanted or indicated for implant with a pacemaker, Implantable Cardioverter-Defibrillator (ICD), Cardiac Resynchronization Therapy (CRT), or hemodynamic monitoring system
* Patient is participating in another clinical study that may have an impact on the study endpoints
* Patient's life expectancy is less than 1 year
* Patient is pregnant
* Patient has unusual thoracic anatomy or scarring at the implant site which may adversely affect the success of the implant procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients recruited for participation in study were indicated for continuous arrhythmia monitoring.
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2010-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reveal In-Office Implants Clinical Research Specialist, Study Chair — Medtronic
Locations (9):
- United States (9):
  - La Jolla, California
  - Miramar, Florida
  - Macon, Georgia
  - Munster, Indiana
  - Takoma Park, Maryland
  - Greensboro, North Carolina
  - Kettering, Ohio
  - Amarillo, Texas
  - San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krahn AD, Klein GJ, Yee R, Takle-Newhouse T, Norris C. Use of an extended monitoring strategy in patients with problematic syncope. Reveal Investigators. Circulation. 1999 Jan 26;99(3):406-10. doi: 10.1161/01.cir.99.3.406. PMID 9918528
- [Background] Solano A, Menozzi C, Maggi R, Donateo P, Bottoni N, Lolli G, Tomasi C, Croci F, Oddone D, Puggioni E, Brignole M. Incidence, diagnostic yield and safety of the implantable loop-recorder to detect the mechanism of syncope in patients with and without structural heart disease. Eur Heart J. 2004 Jul;25(13):1116-9. doi: 10.1016/j.ehj.2004.05.013. PMID 15231369
- [Background] Krahn AD, Klein GJ, Yee R, Skanes AC. Detection of asymptomatic arrhythmias in unexplained syncope. Am Heart J. 2004 Aug;148(2):326-32. doi: 10.1016/j.ahj.2004.01.024. PMID 15309004
- [Background] Moya A, Brignole M, Menozzi C, Garcia-Civera R, Tognarini S, Mont L, Botto G, Giada F, Cornacchia D; International Study on Syncope of Uncertain Etiology (ISSUE) Investigators. Mechanism of syncope in patients with isolated syncope and in patients with tilt-positive syncope. Circulation. 2001 Sep 11;104(11):1261-7. doi: 10.1161/hc3601.095708. PMID 11551877
- [Background] Hancox JG, Venkat AP, Coldiron B, Feldman SR, Williford PM. The safety of office-based surgery: review of recent literature from several disciplines. Arch Dermatol. 2004 Nov;140(11):1379-82. doi: 10.1001/archderm.140.11.1379. PMID 15545548
- [Background] Krahn AD, Klein GJ, Norris C, Yee R. The etiology of syncope in patients with negative tilt table and electrophysiological testing. Circulation. 1995 Oct 1;92(7):1819-24. doi: 10.1161/01.cir.92.7.1819. PMID 7671366
- [Background] Krahn AD, Klein GJ, Yee R, Norris C. Final results from a pilot study with an implantable loop recorder to determine the etiology of syncope in patients with negative noninvasive and invasive testing. Am J Cardiol. 1998 Jul 1;82(1):117-9. doi: 10.1016/s0002-9149(98)00237-9. PMID 9671019
- [Background] Seidl K, Breunung S, Rameken M, Siemon G, Schwacke H, Drogemuller A, Zahn R, Senges J. [Initial experience with an implantable loop recorder in patients with unexplained syncope]. Z Kardiol. 2000 Jan;89(1):43-50. doi: 10.1007/s003920050007. German. PMID 10663916
- [Background] Mieszczanska H, Ibrahim B, Cohen TJ. Initial clinical experience with implantable loop recorders. J Invasive Cardiol. 2001 Dec;13(12):802-4. PMID 11731693
- [Background] Krahn AD, Klein GJ, Fitzpatrick A, Seidl K, Zaidi A, Skanes A, Yee R. Predicting the outcome of patients with unexplained syncope undergoing prolonged monitoring. Pacing Clin Electrophysiol. 2002 Jan;25(1):37-41. doi: 10.1046/j.1460-9592.2002.00037.x. PMID 11877934
- [Background] Armstrong VL, Lawson J, Kamper AM, Newton J, Kenny RA. The use of an implantable loop recorder in the investigation of unexplained syncope in older people. Age Ageing. 2003 Mar;32(2):185-8. doi: 10.1093/ageing/32.2.185. PMID 12615562
- [Background] Sanfins V, Chaves JC, Alves A, Silva F, Machado I, Quelhas I, Medeiros R, Pires R, Reis D, Pereira A, de Almeida J. Use of an implantable loop recorder: initial experience. Rev Port Cardiol. 2003 Dec;22(12):1479-83. English, Portuguese. PMID 15008063
- [Background] Mason PK, Wood MA, Reese DB, Lobban JH, Mitchell MA, DiMarco JP. Usefulness of implantable loop recorders in office-based practice for evaluation of syncope in patients with and without structural heart disease. Am J Cardiol. 2003 Nov 1;92(9):1127-9. doi: 10.1016/j.amjcard.2003.07.011. PMID 14583373
- [Background] Donateo P, Brignole M, Menozzi C, Bottoni N, Alboni P, Dinelli M, Del Rosso A, Croci F, Oddone D, Solano A, Puggioni E. Mechanism of syncope in patients with positive adenosine triphosphate tests. J Am Coll Cardiol. 2003 Jan 1;41(1):93-8. doi: 10.1016/s0735-1097(02)02621-9. PMID 12570950
- [Background] Ermis C, Zhu AX, Pham S, Li JM, Guerrero M, Vrudney A, Hiltner L, Lu F, Sakaguchi S, Lurie KG, Benditt DG. Comparison of automatic and patient-activated arrhythmia recordings by implantable loop recorders in the evaluation of syncope. Am J Cardiol. 2003 Oct 1;92(7):815-9. doi: 10.1016/s0002-9149(03)00889-0. PMID 14516882
- [Background] Paisey JR, Yue AM, Treacher K, Roberts PR, Morgan JM. Implantable loop recorders detect tachyarrhythmias in symptomatic patients with negative electrophysiological studies. Int J Cardiol. 2005 Jan;98(1):35-8. doi: 10.1016/j.ijcard.2003.06.020. PMID 15676163
- [Background] Lombardi F, Calosso E, Mascioli G, Marangoni E, Donato A, Rossi S, Pala M, Foti F, Lunati M. Utility of implantable loop recorder (Reveal Plus) in the diagnosis of unexplained syncope. Europace. 2005 Jan;7(1):19-24. doi: 10.1016/j.eupc.2004.09.003. PMID 15670962
- [Background] Inamdar V, Mehta S, Juang G, Cohen T. The utility of implantable loop recorders for diagnosing unexplained syncope in 100 consecutive patients: five-year, single-center experience. J Invasive Cardiol. 2006 Jul;18(7):313-5. PMID 16816436
- [Background] Maggi R, Menozzi C, Brignole M, Podoleanu C, Iori M, Sutton R, Moya A, Giada F, Orazi S, Grovale N. Cardioinhibitory carotid sinus hypersensitivity predicts an asystolic mechanism of spontaneous neurally mediated syncope. Europace. 2007 Aug;9(8):563-7. doi: 10.1093/europace/eum092. Epub 2007 May 16. PMID 17507364
- [Background] Pakarinen S, Oikarinen L, Toivonen L. Short-term implantation-related complications of cardiac rhythm management device therapy: a retrospective single-centre 1-year survey. Europace. 2010 Jan;12(1):103-8. doi: 10.1093/europace/eup361. PMID 19914920
- [Background] Wiegand UK, LeJeune D, Boguschewski F, Bonnemeier H, Eberhardt F, Schunkert H, Bode F. Pocket hematoma after pacemaker or implantable cardioverter defibrillator surgery: influence of patient morbidity, operation strategy, and perioperative antiplatelet/anticoagulation therapy. Chest. 2004 Oct;126(4):1177-86. doi: 10.1378/chest.126.4.1177. PMID 15486380
- [Background] Al-Khatib SM, Lucas FL, Jollis JG, Malenka DJ, Wennberg DE. The relation between patients' outcomes and the volume of cardioverter-defibrillator implantation procedures performed by physicians treating Medicare beneficiaries. J Am Coll Cardiol. 2005 Oct 18;46(8):1536-40. doi: 10.1016/j.jacc.2005.04.063. Epub 2005 Sep 23. PMID 16226180
- [Background] Chamis AL, Peterson GE, Cabell CH, Corey GR, Sorrentino RA, Greenfield RA, Ryan T, Reller LB, Fowler VG Jr. Staphylococcus aureus bacteremia in patients with permanent pacemakers or implantable cardioverter-defibrillators. Circulation. 2001 Aug 28;104(9):1029-33. doi: 10.1161/hc3401.095097. PMID 11524397
- [Background] Brignole M, Sutton R, Menozzi C, Garcia-Civera R, Moya A, Wieling W, Andresen D, Benditt DG, Vardas P; International Study on Syncope of Uncertain Etiology 2 (ISSUE 2) Group. Early application of an implantable loop recorder allows effective specific therapy in patients with recurrent suspected neurally mediated syncope. Eur Heart J. 2006 May;27(9):1085-92. doi: 10.1093/eurheartj/ehi842. Epub 2006 Mar 28. PMID 16569653
- [Background] Brignole M, Menozzi C, Moya A, Garcia-Civera R, Mont L, Alvarez M, Errazquin F, Beiras J, Bottoni N, Donateo P; International Study on Syncope of Uncertain Etiology (ISSUE) Investigators. Mechanism of syncope in patients with bundle branch block and negative electrophysiological test. Circulation. 2001 Oct 23;104(17):2045-50. doi: 10.1161/hc4201.097837. PMID 11673344
- [Background] Menozzi C, Brignole M, Garcia-Civera R, Moya A, Botto G, Tercedor L, Migliorini R, Navarro X; International Study on Syncope of Uncertain Etiology (ISSUE) Investigators. Mechanism of syncope in patients with heart disease and negative electrophysiologic test. Circulation. 2002 Jun 11;105(23):2741-5. doi: 10.1161/01.cir.0000018125.31973.87. PMID 12057988
- [Background] Vater M., Rameken M., Pitschner H.F., et al. The endless-loop-recorder in clinical practice - Results of the multicentre German Reveal® registry. Herzschrittmachertherapie und Elektrophysiologie (2002) 13:2 (101-109).
- [Derived] Pachulski R, Cockrell J, Solomon H, Yang F, Rogers J. Implant evaluation of an insertable cardiac monitor outside the electrophysiology lab setting. PLoS One. 2013 Aug 15;8(8):e71544. doi: 10.1371/journal.pone.0071544. eCollection 2013. PMID 23977071

RESULTS

PARTICIPANT FLOW:
Groups:
- Enrollment Cohort: Enrollment cohort includes any patients who meet the inclusion and exclusion criteria and have a signed inform consent.
Period: Overall Study
Arm/Group | Enrollment Cohort
Started | 66
Completed | 65
Not Completed | 1
Not completed — Patient exited prior to implant | 1

BASELINE CHARACTERISTICS:
Arm/Group | Enrollment Cohort
Number analyzed (Participants) | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (17.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 36
Region of Enrollment [Number; unit: participants]
  United States | 66

OUTCOME MEASURES:

1. Primary Outcome: Procedure-related Complications Rate Requiring Resolution by Surgical Intervention
Description: This objective estimates the proportion of patients having procedure-related complication requiring resolution by surgical intervention at 90 days post-implant procedure using Kaplan-Meier method.
Time Frame: From Implant to 90 days post-implant procedure
Population: Reveal device indicated patients, enrolled in the study and implanted per protocol
Measure: Number; unit: participants
Groups:
- Implant Cohort: Patient with Reveal device implanted
Arm/Group | Implant Cohort
Number analyzed (Participants) | 65
participants | 2
Statistical Analysis 1: Comparison: Implant Cohort; Test type: Other — There was no formal statistical hypothesis tested. The goal was to estimate the procedure-related complications 90 days post implant using the Kaplan-Meier method; Rate = 0.034, 95% CI 1-sided [upper limit 0.1292]

2. Secondary Outcome: Number of Participants Having Procedure-related Adverse Events
Description: Report number of participants having procedure-related adverse events that meet the primary endpoint (requiring surgical intervention), and number of participants having other procedure-related adverse events (not requiring surgical intervention).
Time Frame: From Implant to 90 days post-implant procedure
Measure: Number; unit: participants
Arm/Group | Implant Cohort
Number analyzed (Participants) | 65
participants
  AEs that meet the primary endpoint | 2
  Other procedure-related AEs | 4

3. Secondary Outcome: Surgical Staff Utilized for Reveal In-office Implants
Description: Observational analysis of surgical staff present at the Reveal Implants
Time Frame: At implant
Reporting Status: Not Posted

4. Secondary Outcome: Techniques and Procedures Utilized During Reveal In-office Implants
Description: Observational data collection as to the technics and procedures utilized during all implants including (but not limited to): device orientation, suturing, wound closure, instrument and material use, and time.
Time Frame: At implant
Reporting Status: Not Posted

5. Secondary Outcome: Physician Satisfaction With Reveal In-office Implants
Description: Observational survey of physicians satisfaction post implant At implant
Time Frame: At implant
Reporting Status: Not Posted

6. Secondary Outcome: R-wave Amplitude Measurement
Description: Average R-wave amplitude at implant and 30-days post procedure
Time Frame: Implant procedure and 30 days post-implant procedure
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From Implant to 90 days post-implant procedure
Arm/Group | Implant Cohort
Serious Adverse Events (participants affected / at risk) | 0/65
Other Adverse Events (participants affected / at risk) | 6/65
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implant Cohort (N=65)
Allergic (Skin and subcutaneous tissue disorders) | 2 (2)
Adverse event require surgical intervention (Infections and infestations) | 2 (2)
Adverse event resolved by oral antibiotics (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No